CLINICAL TRIAL: NCT04855006
Title: Transplantation of Vaginal Mikrobiome - A Randomized, Double-blinded, Controlled Trial
Brief Title: Transplantation of Vaginal Mikrobiome
Acronym: DyscoverII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Henriette Svarre Nielsen, MD, DMSc, Professor, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HH-Dyscover-2021
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Vaginal Dysbiosis; Vaginal Microbiome; Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants are aware if they are allocated as donors or recipients. If the participants are allocated as recipients, they are blinded towards receiving experimental treatment or placebo treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaginal Microbiome Transplant (Experimental): Women are given the vaginal microbiome transplant at least one time and up to three times. If the woman receives the transplant more than once, it will be 28 days after the first transplant and again 28 days after the second transplant.
  Interventions: Biological: Vaginal Microbiome Transplant
- Vaginal Microbiome Transplant Placebo (Placebo Comparator): Women are given the vaginal microbiome transplant placebo at least one time and up to three times. If the woman receives the transplant more than once, it will be 28 days after the first transplant and again 28 days after the second transplant.
  Interventions: Biological: Vaginal Microbiome Transplant Placebo
- Vaginal Microbiome Donors (Experimental): Women allocated in the donor group will donate their vaginal secretion, which will be processed and analyzed throughy before it is used as a transplant. In total, the donors will each provide approximately 10 donations of vaginal secretion.
  Interventions: Other: No intervention

INTERVENTIONS:
Biological: Vaginal Microbiome Transplant — Vaginal Microbiome Transplant is given at least once and up to three times. The transplant is admitted with a syringe
  Arms: Vaginal Microbiome Transplant
Biological: Vaginal Microbiome Transplant Placebo — Vaginal Microbiome Transplant Placebo is given at least once and up to three times. The transplant Placebo is admitted with a syringe
  Arms: Vaginal Microbiome Transplant Placebo
Other: No intervention — Donors have no intervention. This group deliver the transplant to arm 'Vaginal Microbiome Transplant'.
  Arms: Vaginal Microbiome Donors

SUMMARY:
Vaginal dysbiosis is a common condition among women. Vaginal dysbiosis covers imbalances in the vaginal flora, caused by the composition of microbes, bacteria, viruses and fungi. Dysbiosis occurs in about 16% of all women in Denmark. A large proportion of women who have vaginal dysbiosis do not experience any symptoms.

However, vaginal dysbiosis can present challenges in several contexts, including a higher tendency for bacterial infections in the female genitals, lower chances of pregnancy in women undergoing fertility treatment, just as it can predispose to premature birth.

This project is aimed at women aged 18-40, who wants to participate in a study to investigate whether, by transplanting vaginal secretion from one woman with a normal vaginal bacterial flora to another woman with an imbalance in the vaginal bacterial flora (called vaginal dysbiosis), can establish a normal vaginal bacterial flora in the recipient of the transplant.

The study will also explore weather genetic, immunological, hormonal, metabolic, health behaviors and clinical factors have significance on whether a normal vaginal flora is achieved after transplantation.

DETAILED DESCRIPTION:
06.12.2021 - Amendment to protocol. A subgroup of 24 women included in the main study as recipients, were asked to participate in delivery of menstrual blood (2-3 times) and peripheral blood (2-3 times). This to analyse immunological cells via flowcytometry in women with vaginal dysbiosis and if there is a change after engraftment of the VMT product.

17.05.2022 - Amendment to protocol. Those/if any women who did not convert their vaginal microbiome is asked to participate in a substudy with 2 arms. Local pretreatment with antiseptic and saline water before VMT and local pretreatment with saline water before VMT.

26.09.2022 - Amendment to protocol. Study arm with only pretreatment of antiseptic was added to the amendment from the 17.05.2022.

ELIGIBILITY:
Inclusion Criteria:

Donor:

* a woman between 18 and 40 years old;
* generally healthy and do not suffer from an immunological or other chronic diseases;
* have regular menstruation or do not menstruate due to birth control pills, gestagen pills (mini-pills), etonogestrel birth control implant or hormone IUD;
* not or do not have a desire to become pregnant within the next year;
* willing to be asked personal questions in the form of medical history, current use of medication, sexuality and sexual behavior;
* willing to refrain from vaginal intercourse unless a condom is used during certain periods of participation; and
* can read and understand information material in Danish or English.
* Accept not to use any intravaginal products such as tampons, menstrual cup, sex toys, vaginal cleaning products, spermicide products and vaginal lubrication.

Recipient:

* a woman between 18 and 40 years old;
* generally healthy and do not suffer from an immunological or other chronic diseases;
* have regular menstruation or do not menstruate due to birth control pills, gestagen pills (mini-pills), etonogestrel birth control implant or hormone IUD;
* not or do not have a desire to become pregnant within the next year;
* willing to be asked personal questions in the form of medical history, current use of medication, sexuality and sexual behavior;
* willing to refrain from vaginal intercourse unless a condom is used during certain periods of participation; and
* can read and understand information material in Danish or English.
* Accept not to use any intravaginal products such as tampons, menstrual cup, sex toys, vaginal cleaning products, spermicide products and vaginal lubrication.

Exclusion Criteria:

Donor:

* Being pregnant
* Any medical history of bacterial vaginosis, Trichomoniasis, Syphilis, HPV, herpes, intraabdominal infections, recurrent urine infections or Mycoplasma infections.
* Positive test result of HIV, Hepatitis A, B and C, Chlamydia, Gonorré, Mycoplasma, Trichonomas, HPV, herpes simplex and Streptococcus A, B, C and G.
* Currently pregnant or lactating.
* Any history of Gonorré and/or Chlamydia during the last year.
* Have been travelling or have had a sexual partner who has been travelling to countries with Ebola and/or Zika virus within the last year.
* Any other medical history, current use of medicine, travels or behavior which from a doctor's perspective is considered not suitable for being a donor.
* Hysterectomized
* Have participated in other medical studies within the last 30 days
* Removal of IUD, cervical cryotheraphy or cervical laser-treatment up until 3 months before screening.
* Any condition requiring the use of antibiotics in the investigation period
* Usage of long-acting hormonal therapy within the last 3 months prior to screening.
* Any social, medical or psychological condition including any history of drug and alcohol abuse, where it is evaluated that the participant cannot adhere to the protocol
* Unsatisfying examination and screening results evaluated by a doctor
* Any sexual habits, history or sexual partner, where the behavior can lead to an increased risk of sexual infections.
* Usage of medicine, recently vaccinated or other behavior which is considered to be a hinder for participation.

Recipient:

* Being pregnant
* Planning to become pregnant within the next 6 months
* Lactating
* Being less than 8 weeks post partum
* Known positive HIV/AIDS infection or other immune diseases
* Positive test result of HIV, Hepatitis A, B and C, Chlamydia, Gonorré, Mycoplasma, Trichonomas, positive urine hCG and HPV.
* Have participated in other medical studies within the last 30 days
* Removal of IUD, cervical cryotheraphy or cervical laser-treatment up until 3 months before screening.
* Any condition requiring the use of antibiotics in the investigation period
* Usage of long-acting hormonal therapy within the last 3 months prior to screening.
* Any social, medical or psychological condition including any history of drug and alcohol abuse, where it is evaluated that the participant cannot adhere to the protocol
* Unsatisfying examination and screening results evaluated by a doctor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on gender identity.
Enrollment: 302 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Engraftment of transplanted vaginal microbiome | 63 days from transplantation
  The number of patients who shifts from having a vaginal dysbiosis to not having a vaginal dysbiosis 7 days after the transplant - up to 3 transplants.

SECONDARY OUTCOMES:
Engraftment of transplanted vaginal microbiome after one transplantation | 7 days from transplantation
  The number of patients who shifts from having a vaginal dysbiosis to not having a vaginal dysbiosis 7 days after the transplant.
Changes in the recipients vaginal bacterial composition | 63 days from transplantation
  Changes in the recipients vaginal bacterial composition after and during the intervention time

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided